CLINICAL TRIAL: NCT06491719
Title: A Study on Efficacy and Safety of iNK Cell Infusion in Patients With Chronic Active Epstein-Barr Virus Infection (CAEBV) and Epstein Barr Virus-induced Haemophagocytic Lymphohistiocytosis (EBV-HLH) After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Study on Efficacy and Safety of iNK Cells for CAEBV /EBV-HLH After Allo-HSCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-P2-053-02
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: CAEBV (Chronic Active Epstein-Barr Virus Infection) Syndrome; EBV; Hemophagocytic Lymphohistiocytoses
MeSH Terms: conditions — Syndrome; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iNK cells infusion patients (Experimental): Given iNK cell infusion after allo HSCT
  Interventions: Other: NCR300（Allogenic Ipsc-derived Natural Killer cells ）

INTERVENTIONS:
Other: NCR300（Allogenic Ipsc-derived Natural Killer cells ） — Patients will receive iNK cells i.V. infusion at 1.0x10^8/kg on days +14d, +21d, +28d, and +35d post-transplant.
  Continuation of the infusion after +35d post-transplant is at the discretion of the physician based on the patient's benefit.

SUMMARY:
To evaluate the efficacy and safety of iNK cells infusion in patients with chronic active Epstein-Barr virus infection (CAEBV) and EBV-associated hemophagocytic lymphohistiocytosis (EBV-HLH) after allogeneic hematopoietic stem cell transplantation (allo-HSCT)

DETAILED DESCRIPTION:
It is a prospective, open-lable study to evaluate the efficacy and safety of iNK cell infusion in CAEBV/EBV-HLH patients after allo-HSCT. The study will enroll fifteen subjects who will receive ongoing least 4 doses of iNK cells intravenously infusion after allogeneic hematopoietic stem cell transplantation. All subjects will assess the incidence of disease relapse and EBV-DNA reactivation up to one year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CAEBV or EBV-HLH who are eligible for allogeneic hematopoietic stem cell transplantation meet one of the following criteria:

   ①EBV-DNA (PBMC or plasma) was still more than 103 before transplantation；②Positive for Cerebrospinal fluid EBV-DNA；

   ③Abnormal phenotypic lymphocytes could still be detected in bone marrow immunotyping；

   ④Measurable EBV-related lesions on imaging；
2. ≤65 years，ECOG :0-2；
3. Cardiac EF≥40%, creatinine clearance ≥50%; aminotransferase（ALT/AST）<200U/L。；
4. In patients with HLH, HLH efficacy ≥Partial Response after prior treatment is required；
5. Estimated survival time is longer than three months；
6. Agree to sign the Informed Consent Form。

Exclusion Criteria:

1. Patients with evidence of grade II or more serious heart disease according to the New York Heart Association (NYHA) score (including Grade II) ; Clear diagnosis of cirrhosis；
2. Active infections other than EBV that have not yet been controlled；
3. Positive for hepatitis B virus or hepatitis C virus；
4. Active massive hemorrhage of internal organs (including gastrointestinal hemorrhage, alveolar hemorrhage, intracranial hemorrhage, etc.)；
5. Also participation in other interventional clinical studies within 4 weeks

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time (DFS) | 1 year
  Assessment of CAEBV, EBV-HLH systemic disease status and peripheral blood EBV-DNA levels
complete remission rate (CR) | 1 year
  EBV-DNA negative rate in relapsed/non-remitting patients
Recurrence rate (RT) | 1 year
  EBV-DNA reactivation rate for high-risk patients

SECONDARY OUTCOMES:
cytomegalovirus DNA | 1 year
  Incidence of post-transplant infection-related comorbidities
Adverse Event（AE） | 1 year
  Assess the frequency and extent of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No